CLINICAL TRIAL: NCT05297760
Title: Documentation of Efficacy for Intralymphatic Allergen Immunotherapy in a Phase III Randomized, Parallel Group, Double Blind Placebo-controlled Multisite Field Trial
Brief Title: Intralymphatic Immunotherapy With Polvac Grass & Rye Allergen Extract
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Pal Johansen, Professor Dr. sc., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University Hospital Zurich
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rhinitis, Allergic, Seasonal; Rhinitis; Allergic, With Asthma; Allergic Rhinitis; Allergic Rhinitis Due to Grass Pollen; Allergic Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Rhinitis, Allergic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polvac (Active Comparator): Polvac Grass+Rye
  Interventions: Biological: Polvac Grass+Rye
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: Polvac Grass+Rye; Drug: Saline 0.9%

INTERVENTIONS:
Biological: Polvac Grass+Rye — Suspension of micro crystalline tyrosine with grass and rye pollen allergen
  Other Names: Polvac
Drug: Saline 0.9% — Physiological saline solution for use as vehicle for the biological drug (Polvac Grass+Rye) or as placebo.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The primary goal is to investigate the efficacy of intralymphatic immunotherapy (ILIT) for the treatment of allergic rhinitis and allergic asthma due to sensitisation to grass pollen allergens. 60 patients with allergic rhinitis will be included and randomized to receive either Polvac (n=30) or placebo (n=30). All patients will receive three injections with 4-8 weeks interval. The injections into a inguinal lymph node is guided by sonography.

Patients will record symptoms and medication use in the summer of 2022 and 2023.

DETAILED DESCRIPTION:
This study is part of a multicenter trial Phase III that takes place also in Denmark and Sweden (EudraCT registration number 2020-001060-28). The primary goal is to investigate the efficacy of intralymphatic immunotherapy (ILIT) for the treatment of allergic rhinitis and allergic asthma due to sensitisation to grass pollen allergens.

In the Swiss arm of trial, Polvac (Allergy Therapeutics, United Kingdom) is applied. In Denmark and Sweden, the applied drug is Alutard (ALK, Denmark). The major difference is the excipient adjuvant, which is microcrystallin tyrosine (MCT) in Polvac aluminium in Alutard. The concentration of major allergen 60 phl p5, as the active ingredient, is the same in both products. The active ingredient is a standardised grass pollen allergen extract combined with MCT. The allergen extract has been treated with glutaraldehyd as to reduce allergenicity, i.e., increase the safety. In Switzerland and Germany, Bencard AG is providing the product. Polvac™, is a marketed product that is approved by the Swiss Medical Product Agencies and adheres to GMP. The product consists of needle-like crystalline structures of average 20 micrometer size. Polvac is approved for subcutaneous immunotherapy (SCIT), which consists of 6 pre-seasonal injections with 1-2 week intervals for 3-4 years, adding up to a total of 18 to 24 injections for the treatment to be completed.

In the currents study, 60 patients with allergic rhinitis will be included and randomized to receive either Polvac (n=30) or placebo (n=30). Primary screening is done online through questionnaires. Secondary screening and inclusion is done clinical at the University Hospital Zurich. All patients will receive three injections of Polvac or placebo (saline) with 4-8 weeks interval. The injections into a inguinal lymph node is guided by sonography.

For three days post each injections, adverse events will be recorded by patients using an on line application. In the summer seasons of 2022 and of 2023, the patients will record daily allergic symptoms and daily medication usage using an online application. These record are the basics for the efficacy analysis.

Addition on January 12th 2024:

After unblinding of the study in October to December 2023 and after analysis of the primary endpoint, it was decided to prolong the study in a semi-cross over. That means, study participants that received placebo in the original trial (n=30) will receive active treatment in an open label setting. The treatment will be exact similar to that of the active treatment in 2022, i.e., three ILIT injections of the IMD (Polvac Grass+Rye) with 4 weeks intervals and using the same dose as in 2022. The study participants that originally received active treatment (n=30) will not receive further treatment.

All patients (n=60), will be invited to enter symptoms and medication usage during the pollen season of 2024, similar to 2022 and 2023. In September to November 2024, the all patients will be invited for a final follow-up visit for clinical and laboratory tests. All patients will concent to the trial extension in writing prior to entering the trial extension.

ELIGIBILITY:
Inclusion Criteria:

* passed online screening with a Rhinoconjunctivitis Total Symptom Score (RTSS) value of 8 or higher.
* sensitisation to grass pollen allergens with a skin prick test reaction to grass pollen allergen of 3 mm or more.
* eligible to allergen immunotherapy.
* 18 years or older.
* comfortable with digital data entry.

Exclusion Criteria:

* previous grass pollen-specific immunotherapy.
* significant allergy to mugwort or pet animal allergens.
* uncontrolled asthma.
* upper airway disease.
* severe pulmonary disease.
* recent allergic reactions.
* immunosuppression.
* cardiovascular disease.
* malignant disease.
* use of ACE-blockers.
* other diseases or conditions rendering the treatment of anaphylactic reactions difficult.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Combined symptom medication score (cSMS) | 3 months (2 minutes per day)
  Daily registration of symptoms and medication usage by the study participants and by means of a online application. This is done during the pollen season of 2022 (and possible 2023 if the 2022 season is poor with low amounts of pollen). The assessment is done over a time period, but the records are integrated for the calculation of one single score (cSMS), which is the primary outcome.

SECONDARY OUTCOMES:
Rhino conjunctivitis quality of life score (RQLQ) | 3 months (10 minutes per week)
  Weekly questionnaire for studying the quality of life of the study participants during the pollen season of 2022 (and possible 2023 if the 2022 season is poor with low amounts of pollen). The RQLQ will assess seven domains on a weekly basis on a scale from 0 (best) to 6 (worst). The assessment is done over a long time period, but the records are integrated for the calculation of one single score (RQLC), which is the secondary outcome.
Lower airway disease | 10 minutes (5 times in two years)
  We will assess spirometry, at each follow-up time point (winter and summer visits) and analyse a time series of the development of each parameter in each treatment group. The assessments will be performed at several time-points and the changes from baseline assessments (before ILIT) is measured.
Asthma | 10 minutes (5 times in two years)
  We will assess FeNo (Fraction Exspiratory Nitric Oxide) at each follow-up time point (winter and summer visits) and analyse a time series of the development of each parameter in each treatment group. The assessments will be performed at several time-points and the changes from baseline assessments (before ILIT) are measured.
Biomarkers | 5 minutes (8 times in two years)
  Circulating levels of IgE, IgG1, and IgG4 specific for grass pollen extract and the major allergens Phl p 5 and Phl p 1 will be determined in blood samples before every treatment and at all the follow-up visits, for a total of 7 times per participant. The analysis is done using ImmunoCAP ELISA. In addition, IgE assessment by ISAC (112 allergens in one array) will be performed to analyse if sensitisation to other allergens develops or changes. All assessments will be performed at several time-points and the changes from baseline assessments (before ILIT) are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pål Johansen, PhD, Principal Investigator — Univeristät Zürich, Dermatologische Klinik
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Anonymous data can be shared on request by contacting the principle investigator. The shared info can include:
  * Study Protocol
  * Statistical Analysis Plan (SAP)
  * Informed Consent Form (ICF)
  * Clinical Study Report (CSR)

REFERENCES:
- [Result] Senti G, Freiburghaus AU, Larenas-Linnemann D, Hoffmann HJ, Patterson AM, Klimek L, Di Bona D, Pfaar O, Ahlbeck L, Akdis M, Weinfeld D, Contreras-Verduzco FA, Pedroza-Melendez A, Skaarup SH, Lee SM, Cardell LO, Schmid JM, Westin U, Dollner R, Kundig TM. Intralymphatic Immunotherapy: Update and Unmet Needs. Int Arch Allergy Immunol. 2019;178(2):141-149. doi: 10.1159/000493647. Epub 2018 Nov 2. PMID 30391954
- [Result] Freiberger SN, Zehnder M, Gafvelin G, Gronlund H, Kundig TM, Johansen P. IgG4 but no IgG1 antibody production after intralymphatic immunotherapy with recombinant MAT-Feld1 in human. Allergy. 2016 Sep;71(9):1366-70. doi: 10.1111/all.12946. Epub 2016 Jun 17. PMID 27253988
- [Result] Zaleska A, Eiwegger T, Soyer O, van de Veen W, Rhyner C, Soyka MB, Bekpen C, Demiroz D, Treis A, Sollner S, Palomares O, Kwok WW, Rose H, Senti G, Kundig TM, Ozoren N, Jutel M, Akdis CA, Crameri R, Akdis M. Immune regulation by intralymphatic immunotherapy with modular allergen translocation MAT vaccine. Allergy. 2014 Sep;69(9):1162-70. doi: 10.1111/all.12461. Epub 2014 Jul 12. PMID 24934402
- [Result] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Result] Senti G, Johansen P, Kundig TM. Intralymphatic immunotherapy. Curr Opin Allergy Clin Immunol. 2009 Dec;9(6):537-43. doi: 10.1097/ACI.0b013e3283310ff7. PMID 19680119
- [Result] Senti G, Prinz Vavricka BM, Erdmann I, Diaz MI, Markus R, McCormack SJ, Simard JJ, Wuthrich B, Crameri R, Graf N, Johansen P, Kundig TM. Intralymphatic allergen administration renders specific immunotherapy faster and safer: a randomized controlled trial. Proc Natl Acad Sci U S A. 2008 Nov 18;105(46):17908-12. doi: 10.1073/pnas.0803725105. Epub 2008 Nov 10. PMID 19001265
- [Result] Skaarup SH, Schmid JM, Skjold T, Graumann O, Hoffmann HJ. Intralymphatic immunotherapy improves grass pollen allergic rhinoconjunctivitis: A 3-year randomized placebo-controlled trial. J Allergy Clin Immunol. 2021 Mar;147(3):1011-1019. doi: 10.1016/j.jaci.2020.07.002. Epub 2020 Jul 15. PMID 32679209
- [Result] Schmid JM, Nezam H, Madsen HH, Schmitz A, Hoffmann HJ. Intralymphatic immunotherapy induces allergen specific plasmablasts and increases tolerance to skin prick testing in a pilot study. Clin Transl Allergy. 2016 May 25;6:19. doi: 10.1186/s13601-016-0107-x. eCollection 2016. PMID 27231527
- [Result] Skaarup SH, Graumann O, Schmid J, Bjerrum AS, Skjold T, Hoffmann HJ. The number of successful injections associates with improved clinical effect in intralymphatic immunotherapy. Allergy. 2021 Jun;76(6):1859-1861. doi: 10.1111/all.14642. Epub 2020 Nov 16. No abstract available. PMID 33099797
- [Result] Aini NR, Mohd Noor N, Md Daud MK, Wise SK, Abdullah B. Efficacy and safety of intralymphatic immunotherapy in allergic rhinitis: A systematic review and meta-analysis. Clin Transl Allergy. 2021 Aug 17;11(6):e12055. doi: 10.1002/clt2.12055. eCollection 2021 Aug. PMID 34429875
- [Result] Werner MT, Bosso JV. Intralymphatic immunotherapy for allergic rhinitis: A systematic review and meta-analysis. Allergy Asthma Proc. 2021 Jul 1;42(4):283-292. doi: 10.2500/aap.2021.42.210028. PMID 34187620
- [Result] Hoang MP, Seresirikachorn K, Chitsuthipakorn W, Snidvongs K. Intralymphatic immunotherapy for allergic rhinoconjunctivitis: a systematic review and meta-analysis. Rhinology. 2021 Jun 1;59(3):236-244. doi: 10.4193/Rhin20.572. PMID 33647073
- See also: Description of the current multicenter trial and registration platform for patient who would like to attend the trial — https://ilit.nu